CLINICAL TRIAL: NCT00173329
Title: The Quality of Life of Patients With Severe Illnesses
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Other Study IDs: 9461700615; NSC93-2314-B-002-294
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-10-21 (Estimated); Status verified 2005-09

CONDITIONS: Schizophrenia; HIV Infections
Keywords: HIV
MeSH Terms: conditions — Schizophrenia; HIV Infections

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Lately researchers and clinicians have emphasized the health related quality of life. Several reasons account for this trend. First of all, the advanced medical practices have contributed to the increased life expectancy. Secondly, the pattern of diseases has shifted from high acuity to chronicity. Therefore, the effectiveness of health care could not be solely evaluated by the rates of morbidity and mortality. The state of patients' quality of life has become the pivotal indicator of the effectiveness of health care interventions. On the other hand, patients' subjective perceptions of health care are crucial factors in treatment processes. Therefore quality of life becomes reference in choosing health care interventions to enhance the benefits of patients.

The scopes of quality of life research include the essence of quality of life, the measurements of quality of life and the relationships between quality of life and its related factors, etc. The local researchers have long put efforts in quality of life research. The results of these studies have contributed to the understandings of different patients' quality of life. However, the majority of studies have focused on specific diseases. This study propose to extend the scope of quality of life research to study patients' quality of life of two severe illnesses, i.e. HIV infections and schizophrenia. These two illnesses represent two severe physical and psychiatric illnesses. Even their etiology, mechanisms, disease process, signs and symptoms, and treatments are different. However, the similarities of these two illnesses include both are severe illnesses without cure, both are stigmatized by the society. Patients with these two illnesses suffer in their personal lives, social relations and quality of life. Therefore the current study to further investigate and compare and contrast the essence of patients' quality of life and their related factors.

The proposed study is a second year study of the two-year study - The quality of life of patients with severe illnesses (NSC93-2314-B-002-294). The first year study focused on the investigation of the quality of life of patients with HIV infections (NSC93-2314-B-002-294). The aim of this proposed study is to compare and contrast the quality of life and its related factors of patients with schizophrenia and HIV infections. The contributions of this study include the in-depth understandings of quality of life of patients with HIV infections and schizophrenia and the comparison of quality of life of different illnesses. The results serve as the foundations in future development of intervention programs to enhance patients' quality of life and cost-effectiveness analyses.

ELIGIBILITY:
Inclusion Criteria:

* people with schizophrenia
* people with HIV

Exclusion Criteria:

-

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2005-08; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Chuan Hsiung, PH.D, Study Chair — National Taiwan University Hospital
Locations (1):
- Ping-Chuan,Hsiung, Taipei, Taiwan